CLINICAL TRIAL: NCT05085223
Title: Development of Hypernatremia in Critically Ill Patients: Prospective Analysis
Brief Title: Prospective Analysis Into Development of Hypernatremia in Critically Ill Patients
Acronym: HYPNIC II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Eveline Mestrom, Principal Investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: HYPNIC II
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Hypernatremia; Critical Illness
MeSH Terms: conditions — Hypernatremia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Daily urine collection for biochemical analysis — For every patient in ICU, a daily morning urine sample will be collected from the already collected urine via catheter.
Other: Subanalysis for comparison of 24hour urine collection versus spot-check measurements — For a subgroup of 30 sedated patients, 24 hour urine collection will be collected. In addition, every 2 hours a 10ml urine sample will be collected.

SUMMARY:
Hypernatremia is frequently encountered in patients admitted to the Intensive Care Unit (ICU) and associated with increased mortality and length of stay. Previous studies focused on predictors in the development and recovery of hypernatremia by including amount and types of administered medication, fluid balance, laboratory results and changes in vital signs. However, data of larger populations or data on infusion rates, fluid and sodium balance or renal replacement therapy is lacking. The predecessor of this study was the HYPNIC trial which found that increased sodium load en decreased sodium excretion preceded hypernatremia development, but was lacking information on the first 48 hours, fluid balances were manually collected before a new data collection system was introduced and was suffering from substantial amounts of missing data and small population for trend analysis.

This study aims to provide better insight in the development and recovery of hypernatremia while paying attention to the limitations from the HYPNIC trial.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Intensive Care Unit
* Age 18 years or older

Exclusion Criteria:

* Age 17 years or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Hypernatremia | During admission in ICU
  After one year of collecting data on fluid and sodium balances, the patients who developed hypernatremia during their admission in the Intensive Care Unit will be compared to the patients who remained normonatremic throughout their ICU admission.

SECONDARY OUTCOMES:
24 hour urine replacement for spot-checks | 24 hours
  Assessing whether 24 hour urine collection can be replaced by spot-check measurements of urine by comparing both 24 hour urine and 2 hourly urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mestrom EHJ, van der Stam JA, Te Pas ME, van der Hoeven JG, van Riel NAW, Bindels AJGH, Boer A, Scharnhorst V. Increased sodium intake and decreased sodium excretion in ICU-acquired hypernatremia: A prospective cohort study. J Crit Care. 2021 Jun;63:68-75. doi: 10.1016/j.jcrc.2021.02.002. Epub 2021 Feb 10. PMID 33621892